CLINICAL TRIAL: NCT06806475
Title: SUSTAINED KETAMINE EFFECTIVENESS for SUICIDAL IDEATION
Acronym: SKESI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Principal Investigator, Emilie OLIE, MD PhD, University Hospital, Montpellier
Other Study IDs: 23.11.07
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2023-11

CONDITIONS: Depression - Major Depressive Disorder; Suicide
Keywords: suicide; depression; major depressive disorder; ketamine
MeSH Terms: conditions — Suicide; Depression; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
As part of the usual clinical activity of the Emergency and Post-Emergency Psychiatric Department, IV ketamine is used to treat suicidal crises in depressed patients hospitalized as an add-on to the treatment of depression. This infusion can be repeated.

Patients are systematically reassessed twice in the month following the last infusion, to ensure that the suicidal crisis is progressing. Psychometric assessments are part of routine care, to ensure systematic evaluation of psychopathology, intensity of depression and suicidality.

Therefore existing data were re-used from the medical records of patients who had received ketamine infusions to assess the effect of ketamine on suicidal ideation and behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with IV ketamine in the Psychiatric Emergency and Post-Emergency Department (University Hospital, Montpellier) in context of suicidal crisis
* over 18 y.o

Exclusion Criteria:

* Opposition to data use
* Subject deprived of liberty (by judicial or administrative decision)
* Subject protected by law (guardianship or curatorship)
* Subject not affiliated to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with IV ketamine in the Psychiatric Emergency and Post-Emergency Department (University Hospital, Montpellier) in context of suicidal crisis over the period from June 2022 to March 2024
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
suicidal ideation at 7 days after IV ketamine administration | 7 days
  evolution of suicidal ideation at 7 days after IV ketamine administration in the context of a suicidal crisis using severity of suicidal ideation according to C-SSRS (COLUMBIA-SUICIDE SEVERITY RATING SCALE)
  The ideation severity subscale ranges from 1 to 5 (higher score indicating more severe ideation). The ideation intensity subscale includes 5 questions each ranging from 1 to 5 (higher score indication more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.

SECONDARY OUTCOMES:
suicidal ideation at 1 month after IV ketamine administration | 1 month
  evolution of suicidal ideation at 7 days after IV ketamine administration in the context of a suicidal crisis using severity of suicidal ideation according to C-SSRS (COLUMBIA-SUICIDE SEVERITY RATING SCALE)
  The ideation severity subscale ranges from 1 to 5 (higher score indicating more severe ideation). The ideation intensity subscale includes 5 questions each ranging from 1 to 5 (higher score indication more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.
Severity of depressive symptomatology at 7 days | 7 days
  change in depressive symptomatology at 1 week using Montgomery-Åsberg Depression Rating Scale (MADRS)
  The scale consists of 10 items rated from 0 to 6. A score between 0 and 6 indicates euthymia, a score between 7 and 19 mild depression, a score between 20 and 34 moderate depression and a score above 34 severe depression.
Severity of depressive symptomatology at 1 month | 1 month
  change in depressive symptomatology at 1 week using Montgomery-Åsberg Depression Rating Scale (MADRS)
  The scale consists of 10 items rated from 0 to 6. A score between 0 and 6 indicates euthymia, a score between 7 and 19 mild depression, a score between 20 and 34 moderate depression and a score above 34 severe depression.
suicidal ideation at 7 days after IV ketamine | 7 days
  number of hospitalization or ER visit for suicidal ideation
suicidal behavior at 1 month after IV ketamine | 1 month
  number of suicide attempts (confirmed, aborted, interrupted)
suicidal behavior at 3 months after IV ketamine | 3 months
  number of suicide attempts (confirmed, aborted, interrupted)
suicidal ideation at 1 month after IV ketamine | 1 month
  number of hospitalization or ER visit for suicidal ideation
suicidal ideation at 3 months after IV ketamine | 3 months
  number of hospitalization or ER visit for suicidal ideation

CONTACTS AND LOCATIONS:
Overall Officials: Emilie OLIE, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital, Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pastre M, Chancel R, Malestroit M, Courtet P, Olie E. Early Response to Ketamine for Suicidal Crisis Reduces Suicidal Events at 3 Months. J Clin Psychiatry. 2025 Jul 23;86(3):25m15829. doi: 10.4088/JCP.25m15829. PMID 40767760